CLINICAL TRIAL: NCT01832441
Title: Study Safety and Efficacy of Bone Marrow Derived Autologous Cells for the Treatment of Diabetes Mellitus. It is Self Funded (Patients' Own Funding) Clinical Trial
Brief Title: Study Safety and Efficacy of Bone Marrow Derived Autologous Cells for the Treatment of Diabetes Mellitus.
Acronym: BMACD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chaitanya Hospital, Pune (Other)
Responsible Party: Principal Investigator, Dr. Sachin Jamadar, CO-Investigator, Chaitanya Hospital, Pune
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00108
Record Dates: First submitted 2013-04-09; First posted 2013-04-16 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Diabetes Mellitus.
Keywords: Diabetes Mellitus stem cells [MNCS ]
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Transfer of autologous MNC intrathecally (Other): single arm Intra thecal transplantation of autologous MNC
  Interventions: Other: Intra thecal transplantation of autologous MNC

INTERVENTIONS:
Other: Intra thecal transplantation of autologous MNC — Intra thecal inj.of 100 millions MNC in 3 doses at 7 days interval

SUMMARY:
This study is Single arm, Single Centre trial to check the Safety and Efficacy of Bone Marrow Derived Autologous mono nuclear cells (100 Million per dose).trial to be conducted for 36 months in patients with diabetes Mellitus in India,Primary outcome measure are abolition or reduction of insulin by>50 percentage by the end of 6 months of ABMSCT-Any reduction in requirement of Insulin dosage and Improvement in HbA1C Level.

DETAILED DESCRIPTION:
his study is Single arm, Single Centre trial to check the Safety and Efficacy of Bone Marrow Derived Autologous mono nuclear cells (100 Million per dose).trial to be conducted for 36 months in patients with diabetes Mellitus in India,Primary outcome measure are abolition or reduction of insulin by>50 percentage by the end of 6 months of ABMSCT-Any reduction in requirement of Insulin dosage and Improvement in HbA1C Level.

ELIGIBILITY:
Inclusion Criteria:

* Patient should suffer from Diabetes Mellitus.
* Willingness to undergo Bone Marrow derived Autologous cell Therapy.
* Ability to comprehend the explained protocol and thereafter give an informed consent as well as sign the required Informed Consent form(ICF) for the study.
* Ability and willingness to regular visit to hospital for protocol procedures and follow up

Exclusion Criteria:

* Patient with History of Immunodeficiency HIV+,Hepatitis B ,HBV and History of Life threatening allergic or immune -Mediated Reaction. the site of bone marrow aspiration potentially limiting Procedure. Alcohol and drug abuse / dependence. Patients with History of Hypertension and Hypersensitive.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-09; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Abolition or reduction of insulin by >50 percentage | 6 months
  - Abolition or reduction of insulin by >50 percentage of ABMSCT by 6 month

SECONDARY OUTCOMES:
Improvement in HbA1C levels | 6 months
  Improvement in HbA1C levels as compared to baseline by the end of 6 months .

CONTACTS AND LOCATIONS:
Overall Officials: ANANT E BAGUL, M.S, Principal Investigator — CHAITANYA HOSPITAL
Locations (1):
- Chaitanya Hospital, Pune, Maharashtra, India